CLINICAL TRIAL: NCT01475357
Title: Intestinal Function in Neonates With Complex Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Sinai Zyblewski, Assistant Professor, Pediatric Cardiology, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR 20394
Record Dates: First submitted 2011-10-06; First posted 2011-11-21 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Congenital Heart Defects; Growth Failure
Keywords: congenital heart defects; growth failure
MeSH Terms: conditions — Heart Defects, Congenital; Failure to Thrive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: NPO pre-operative (Other): 1) Current care - NPO (nothing by mouth) postnatal intestinal function of neonates with complex CHD who receive enteral trophic breastmilk (10cc/kg/day) feeds (intervention) vs NPO (nothing by mouth) in the pre-operative period.
  Interventions: Other: Arm 1: NPO by mouth pre-operative
- Arm 2: Fresh Breast Milk pre-operative (Active Comparator): 2) Intervention - Trophic mother's own fresh (non-frozen) breastmilk gavage feeds via nasogastric tube every 3 hours at 10 cc/kg/day
  Interventions: Other: Arm 2: Fresh Breast Milk pre-operative

INTERVENTIONS:
Other: Arm 1: NPO by mouth pre-operative — Current treatment for infants born with cardiac defects awaiting surgery is to keep them NPO pre-operatively. Arm 1 will make no changes to this current policy.
  Arms: Arm 1: NPO pre-operative
Other: Arm 2: Fresh Breast Milk pre-operative — Infants randomized to Arm 2 of the study will receive their mother's own breast milk pre-operatively.
  Arms: Arm 2: Fresh Breast Milk pre-operative

SUMMARY:
Postnatal intestinal function in cardiac infants. The overall goal of this proposal is to address a widespread health problem in the pediatric cardiac infant population - poor postnatal growth - through a collaborative effort between pediatric cardiology, cardiothoracic surgery, neonatology, microbiology, and immunology. The hypothesis is that term neonates with complex congenital heart disease (CHD) who receive trophic breastmilk feeds in the pre-operative period will show improved gut function than neonates who were strictly NPO (nothing by mouth) in the pre-operative period.

DETAILED DESCRIPTION:
The overall goal of this proposal is to address a widespread health problem in the pediatric cardiac infant population - poor postnatal growth - through a collaborative effort between pediatric cardiology, cardiothoracic surgery, neonatology, microbiology, and immunology. The foundational hypothesis of this proposal is that term neonates (≥ 37 weeks gestation) with complex congenital heart disease (CHD) are vulnerable to disturbances in intestinal mucosal function, permeability, microflora, and local immune function, which ultimately result in feeding intolerance and poor somatic growth. By identifying biologic targets for perioperative intestinal protection, this project has the potential to shift and improve the paradigm of perioperative care for neonates with complex CHD. This pilot study will generate the data necessary to pursue K23 and R01 funding to further investigate postnatal intestinal maturation and function in neonates with complex CHD and cyanosis, specifically as it pertains to local immune function and inflammatory response.

The objectives of this proposal are to perform a single-center (MUSC), prospective, randomized pilot trial to investigate postnatal intestinal function in cardiac infants through the following Specific Aims:

Specific Aim 1: To compare the decrease in intestinal permeability as determined by urine lactulose: mannitol ratios of the trophic breastmilk fed group (intervention) vs. NPO (nothing by mouth) group (current care) amongst neonates with complex CHD over 3 different time points (postnatal day 3-4, post-operative day 7-8, and post-operative day 13-14).

H1: Infants who receive trophic breastmilk feeds in the pre-operative period will demonstrate a more rapid decrease in intestinal permeability (improved postnatal intestinal maturation) over the first 2 weeks of life compared to those infants who were strictly NPO in the pre-operative period.

Specific Aim 2: To compare the duration (in days) until goal enteral feeds are successfully achieved in the trophic breastmilk fed group vs. NPO group.

H1: Infants who receive trophic breastmilk feeds in the pre-operative period will successfully achieve goal enteral feeds in a shorter duration of time compared to those infants who were strictly NPO in the pre-operative period.

Specific Aim 3: To qualitatively compare the intestinal microflora pattern over the first postpartum month as determined by stool microbiota of the trophic breastmilk fed group vs. NPO group.

H1: The microbiota patterns of those infants who receive trophic breastmilk feeds in the pre-operative period will differ from those infants who were strictly NPO in the pre-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects will be male and female neonates admitted to MUSC PCICU or NICU prior to 72 hours of life who are gestational age ≥ 37 weeks.
* inpatient status at MUSC for a minimum of 48 hours prior to planned surgery and have a postnatal diagnosis of complex congenital heart disease - defined as a structural heart defect requiring cardiac surgery (reparative or palliative) prior to hospital discharge.

Exclusion Criteria:

* Infants with hemodynamic instability in the pre-operative period requiring mechanical circulatory support or
* who have the presence of lactate > 3 after the first 24 hours of admission
* admission from home
* major congenital extracardiac abnormalities (i.e. renal, brain, GI)
* cardiac surgery will not be performed at MUSC, and
* mother does not plan to pump breastmilk during the infant's first week of life.

Ages: 37 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2011-10; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in urine lactulose/mannitol ratio over time | post-natal day 3-4 (baseline), post-op days 7 and 14
  Specific Aim 1: compare decrease in intestinal permeability by urine lactulose: mannitol ratios of the trophic breastmilk fed group (intervention) vs. NPO (nothing by mouth) group (current care) amongst neonates with complex CHD over 3 different time points (postnatal day 3-4, post-operative day 7-8, and post-operative day 13-14).

SECONDARY OUTCOMES:
Enteral Feeds | Duration (in days) until goal enteral feeds are achieved, an expected average of 3 weeks
  Specific Aim 2: To compare the duration (in days) until goal enteral feeds are successfully achieved in the trophic breastmilk fed group vs. NPO group.
  H1: Infants who receive trophic breastmilk feeds in the pre-operative period will successfully achieve goal enteral feeds in a shorter duration of time compared to those infants who were strictly NPO in the pre-operative period.
Intestinal Microflora Pattern | 30 days 1st post-partum month
  Specific Aim 3: To qualitatively compare the intestinal microflora pattern over the first postpartum month as determined by stool microbiota of the trophic breastmilk fed group vs. NPO group.
  H1: The microbiota patterns of those infants who receive trophic breastmilk feeds in the pre-operative period will differ from those infants who were strictly NPO in the pre-operative period.

CONTACTS AND LOCATIONS:
Overall Officials: Sinai C Zyblewski, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Anderson JB, Beekman RH 3rd, Border WL, Kalkwarf HJ, Khoury PR, Uzark K, Eghtesady P, Marino BS. Lower weight-for-age z score adversely affects hospital length of stay after the bidirectional Glenn procedure in 100 infants with a single ventricle. J Thorac Cardiovasc Surg. 2009 Aug;138(2):397-404.e1. doi: 10.1016/j.jtcvs.2009.02.033. Epub 2009 May 23. PMID 19619784
- [Background] Kelleher DK, Laussen P, Teixeira-Pinto A, Duggan C. Growth and correlates of nutritional status among infants with hypoplastic left heart syndrome (HLHS) after stage 1 Norwood procedure. Nutrition. 2006 Mar;22(3):237-44. doi: 10.1016/j.nut.2005.06.008. PMID 16500550
- [Background] MEHRIZI A, DRASH A. Growth disturbance in congenital heart disease. J Pediatr. 1962 Sep;61:418-29. doi: 10.1016/s0022-3476(62)80373-4. No abstract available. PMID 14472142
- [Background] Owens JL, Musa N. Nutrition support after neonatal cardiac surgery. Nutr Clin Pract. 2009 Apr-May;24(2):242-9. doi: 10.1177/0884533609332086. PMID 19321898
- [Background] Schwalbe-Terilli CR, Hartman DH, Nagle ML, Gallagher PR, Ittenbach RF, Burnham NB, Gaynor JW, Ravishankar C. Enteral feeding and caloric intake in neonates after cardiac surgery. Am J Crit Care. 2009 Jan;18(1):52-7. doi: 10.4037/ajcc2009405. PMID 19116405
- [Background] Jeffries HE, Wells WJ, Starnes VA, Wetzel RC, Moromisato DY. Gastrointestinal morbidity after Norwood palliation for hypoplastic left heart syndrome. Ann Thorac Surg. 2006 Mar;81(3):982-7. doi: 10.1016/j.athoracsur.2005.09.001. PMID 16488706
- [Background] Pickard SS, Feinstein JA, Popat RA, Huang L, Dutta S. Short- and long-term outcomes of necrotizing enterocolitis in infants with congenital heart disease. Pediatrics. 2009 May;123(5):e901-6. doi: 10.1542/peds.2008-3216. PMID 19403484
- [Background] del Castillo SL, Moromisato DY, Dorey F, Ludwick J, Starnes VA, Wells WJ, Jeffries HE, Wong PC. Mesenteric blood flow velocities in the newborn with single-ventricle physiology: modified Blalock-Taussig shunt versus right ventricle-pulmonary artery conduit. Pediatr Crit Care Med. 2006 Mar;7(2):132-7. doi: 10.1097/01.PCC.0000200999.89777.92. PMID 16474253
- [Background] Harrison AM, Davis S, Reid JR, Morrison SC, Arrigain S, Connor JT, Temple ME. Neonates with hypoplastic left heart syndrome have ultrasound evidence of abnormal superior mesenteric artery perfusion before and after modified Norwood procedure. Pediatr Crit Care Med. 2005 Jul;6(4):445-7. doi: 10.1097/01.PCC.0000163674.53466.CA. PMID 15982432
- [Background] McElhinney DB, Hedrick HL, Bush DM, Pereira GR, Stafford PW, Gaynor JW, Spray TL, Wernovsky G. Necrotizing enterocolitis in neonates with congenital heart disease: risk factors and outcomes. Pediatrics. 2000 Nov;106(5):1080-7. doi: 10.1542/peds.106.5.1080. PMID 11061778
- [Background] Bernstein D, Bell JG, Kwong L, Castillo RO. Alterations in postnatal intestinal function during chronic hypoxemia. Pediatr Res. 1992 Mar;31(3):234-8. doi: 10.1203/00006450-199203000-00008. PMID 1561008
- [Background] Willis L, Thureen P, Kaufman J, Wymore E, Skillman H, da Cruz E. Enteral feeding in prostaglandin-dependent neonates: is it a safe practice? J Pediatr. 2008 Dec;153(6):867-9. doi: 10.1016/j.jpeds.2008.04.074. PMID 19014824
- [Background] Braudis NJ, Curley MA, Beaupre K, Thomas KC, Hardiman G, Laussen P, Gauvreau K, Thiagarajan RR. Enteral feeding algorithm for infants with hypoplastic left heart syndrome poststage I palliation. Pediatr Crit Care Med. 2009 Jul;10(4):460-6. doi: 10.1097/PCC.0b013e318198b167. PMID 19307819
- [Background] del Castillo SL, McCulley ME, Khemani RG, Jeffries HE, Thomas DW, Peregrine J, Wells WJ, Starnes VA, Moromisato DY. Reducing the incidence of necrotizing enterocolitis in neonates with hypoplastic left heart syndrome with the introduction of an enteral feed protocol. Pediatr Crit Care Med. 2010 May;11(3):373-7. doi: 10.1097/PCC.0b013e3181c01475. PMID 19838139
- [Background] Natarajan G, Reddy Anne S, Aggarwal S. Enteral feeding of neonates with congenital heart disease. Neonatology. 2010;98(4):330-6. doi: 10.1159/000285706. Epub 2010 May 7. PMID 20453528
- [Background] Johnson BA, Mussatto K, Uhing MR, Zimmerman H, Tweddell J, Ghanayem N. Variability in the preoperative management of infants with hypoplastic left heart syndrome. Pediatr Cardiol. 2008 May;29(3):515-20. doi: 10.1007/s00246-007-9022-1. Epub 2007 Nov 22. PMID 18034198
- [Background] Bines JE, Walker WA. Growth factors and the development of neonatal host defense. Adv Exp Med Biol. 1991;310:31-9. doi: 10.1007/978-1-4615-3838-7_3. No abstract available. PMID 1809006
- [Background] Walker WA. Role of nutrients and bacterial colonization in the development of intestinal host defense. J Pediatr Gastroenterol Nutr. 2000;30 Suppl 2:S2-7. PMID 10749395
- [Background] Walker WA. The dynamic effects of breastfeeding on intestinal development and host defense. Adv Exp Med Biol. 2004;554:155-70. doi: 10.1007/978-1-4757-4242-8_15. PMID 15384575
- [Background] Fanaro S, Chierici R, Guerrini P, Vigi V. Intestinal microflora in early infancy: composition and development. Acta Paediatr Suppl. 2003 Sep;91(441):48-55. doi: 10.1111/j.1651-2227.2003.tb00646.x. PMID 14599042
- [Background] Penders J, Thijs C, Vink C, Stelma FF, Snijders B, Kummeling I, van den Brandt PA, Stobberingh EE. Factors influencing the composition of the intestinal microbiota in early infancy. Pediatrics. 2006 Aug;118(2):511-21. doi: 10.1542/peds.2005-2824. PMID 16882802
- [Background] Tanaka S, Kobayashi T, Songjinda P, Tateyama A, Tsubouchi M, Kiyohara C, Shirakawa T, Sonomoto K, Nakayama J. Influence of antibiotic exposure in the early postnatal period on the development of intestinal microbiota. FEMS Immunol Med Microbiol. 2009 Jun;56(1):80-7. doi: 10.1111/j.1574-695X.2009.00553.x. Epub 2009 Apr 6. PMID 19385995
- [Background] Goldman AS. The immune system in human milk and the developing infant. Breastfeed Med. 2007 Dec;2(4):195-204. doi: 10.1089/bfm.2007.0024. PMID 18081456
- [Background] Pietz J, Achanti B, Lilien L, Stepka EC, Mehta SK. Prevention of necrotizing enterocolitis in preterm infants: a 20-year experience. Pediatrics. 2007 Jan;119(1):e164-70. doi: 10.1542/peds.2006-0521. Epub 2006 Dec 4. PMID 17145901
- [Background] Raiten DJ, Kalhan SC, Hay WW Jr. Maternal nutrition and optimal infant feeding practices: executive summary. Am J Clin Nutr. 2007 Feb;85(2):577S-583S. doi: 10.1093/ajcn/85.2.577S. PMID 17284759
- [Background] Klagsbrun M. Nutrition Classics. Proceedings of the National Academy of Sciences of the United States of America, October 1978, Volume 75, Number 10: Human milk stimulates DNA synthesis and cellular proliferation in cultured fibroblasts. By Michael Klagsbrun. Nutr Rev. 1988 Jan;46(1):21-3. doi: 10.1111/j.1753-4887.1988.tb05349.x. No abstract available. PMID 3277090
- [Background] Clark JA, Doelle SM, Halpern MD, Saunders TA, Holubec H, Dvorak K, Boitano SA, Dvorak B. Intestinal barrier failure during experimental necrotizing enterocolitis: protective effect of EGF treatment. Am J Physiol Gastrointest Liver Physiol. 2006 Nov;291(5):G938-49. doi: 10.1152/ajpgi.00090.2006. Epub 2006 Jun 22. PMID 16798726
- [Background] Clark JA, Lane RH, Maclennan NK, Holubec H, Dvorakova K, Halpern MD, Williams CS, Payne CM, Dvorak B. Epidermal growth factor reduces intestinal apoptosis in an experimental model of necrotizing enterocolitis. Am J Physiol Gastrointest Liver Physiol. 2005 Apr;288(4):G755-62. doi: 10.1152/ajpgi.00172.2004. Epub 2004 Nov 4. PMID 15528252
- [Background] Dvorak B. Milk epidermal growth factor and gut protection. J Pediatr. 2010 Feb;156(2 Suppl):S31-5. doi: 10.1016/j.jpeds.2009.11.018. PMID 20105663
- [Background] Taylor SN, Basile LA, Ebeling M, Wagner CL. Intestinal permeability in preterm infants by feeding type: mother's milk versus formula. Breastfeed Med. 2009 Mar;4(1):11-5. doi: 10.1089/bfm.2008.0114. PMID 19196035
- [Background] Garofalo RP, Goldman AS. Cytokines, chemokines, and colony-stimulating factors in human milk: the 1997 update. Biol Neonate. 1998;74(2):134-42. doi: 10.1159/000014019. PMID 9691155
- [Background] Hanson LA, Ahlstedt S, Andersson B, Carlsson B, Fallstrom SP, Mellander L, Porras O, Soderstrom T, Eden CS. Protective factors in milk and the development of the immune system. Pediatrics. 1985 Jan;75(1 Pt 2):172-6. PMID 3880886
- [Background] Xanthou M, Bines J, Walker WA. Human milk and intestinal host defense in newborns: an update. Adv Pediatr. 1995;42:171-208. PMID 8540428
- [Background] van Elburg RM, Fetter WP, Bunkers CM, Heymans HS. Intestinal permeability in relation to birth weight and gestational and postnatal age. Arch Dis Child Fetal Neonatal Ed. 2003 Jan;88(1):F52-5. doi: 10.1136/fn.88.1.f52. PMID 12496227
- [Background] Catassi C, Bonucci A, Coppa GV, Carlucci A, Giorgi PL. Intestinal permeability changes during the first month: effect of natural versus artificial feeding. J Pediatr Gastroenterol Nutr. 1995 Nov;21(4):383-6. doi: 10.1097/00005176-199511000-00003. PMID 8583288
- [Background] Weaver LT, Laker MF, Nelson R, Lucas A. Milk feeding and changes in intestinal permeability and morphology in the newborn. J Pediatr Gastroenterol Nutr. 1987 May-Jun;6(3):351-8. doi: 10.1097/00005176-198705000-00008. PMID 3123630
- [Background] He F, Morita H, Ouwehand AC, Hosoda M, Hiramatsu M, Kurisaki J, Isolauri E, Benno Y, Salminen S. Stimulation of the secretion of pro-inflammatory cytokines by Bifidobacterium strains. Microbiol Immunol. 2002;46(11):781-5. doi: 10.1111/j.1348-0421.2002.tb02765.x. PMID 12516776
- [Background] Walsh MC, Kliegman RM. Necrotizing enterocolitis: treatment based on staging criteria. Pediatr Clin North Am. 1986 Feb;33(1):179-201. doi: 10.1016/s0031-3955(16)34975-6. PMID 3081865
- [Background] Weaver LT, Laker MF, Nelson R. Intestinal permeability in the newborn. Arch Dis Child. 1984 Mar;59(3):236-41. doi: 10.1136/adc.59.3.236. PMID 6424583
- [Background] Dvorak B, Khailova L, Clark JA, Hosseini DM, Arganbright KM, Reynolds CA, Halpern MD. Comparison of epidermal growth factor and heparin-binding epidermal growth factor-like growth factor for prevention of experimental necrotizing enterocolitis. J Pediatr Gastroenterol Nutr. 2008 Jul;47(1):11-8. doi: 10.1097/MPG.0b013e3181788618. PMID 18607263
- [Derived] Zyblewski SC, Nietert PJ, Graham EM, Taylor SN, Atz AM, Wagner CL. Randomized Clinical Trial of Preoperative Feeding to Evaluate Intestinal Barrier Function in Neonates Requiring Cardiac Surgery. J Pediatr. 2015 Jul;167(1):47-51.e1. doi: 10.1016/j.jpeds.2015.04.035. Epub 2015 May 8. PMID 25962930